CLINICAL TRIAL: NCT01261884
Title: Exercise Intervention in Pregnancy for Reduction of Blood Pressure in Obese Gravidas
Brief Title: Exercise in Pregnancy for Reduction of Blood Pressure in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Richard S. Legro, M.D., Professor, Obstetrics and Gynecology and Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 33905
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Hypertension; Pregnancy; Preeclampsia; Exercise
Keywords: Pregnancy; Exercise; Hypertension; Preeclampsia; Resistance exercise
MeSH Terms: conditions — Hypertension; Pre-Eclampsia; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Routine prenatal care (No Intervention)
- Exercise support (Experimental)
  Interventions: Behavioral: Exercise support
- Exercise intervention (Experimental)
  Interventions: Behavioral: Exercise intervention

INTERVENTIONS:
Behavioral: Exercise support — Group B (exercise support) will be given the ACOG pamphlet on exercise in pregnancy, a daily activity log, and a pedometer. This group will be asked to wear the pedometer for 7 consecutive days between Visits 1 and 2, and record daily activities.
  Arms: Exercise support
Behavioral: Exercise intervention — Group C (exercise intervention) will be given the ACOG pamphlet on exercise in pregnancy, a daily activity log, a pedometer, a resistance band, and a handout on specific exercises (type and frequency) to be performed. The study coordinator will demonstrate each exercise and then observe the participant perform each exercise to assure full understanding. In addition to wearing the pedometer for 7 days and completing the activity log, this group will also record compliance with the exercise regimen.
  Arms: Exercise intervention

SUMMARY:
Preeclampsia and other high blood pressure disorders of pregnancy are a significant cause of both maternal and fetal complications of pregnancy. To date, there is no known "cure" for preeclampsia, but studies have shown that exercise may lower the risk of preeclampsia and high blood pressure disorders in pregnancy. Resistance training also lowers blood pressure, and may be easier to perform in a pregnant population, leading to higher compliance. The investigators propose to perform a novel prospective study of a resistance training regimen on blood pressure in pregnant patients at high risk for developing preeclampsia or high blood pressure.

DETAILED DESCRIPTION:
Hypertension affects 5-10 percent of pregnancies, and complications from hypertensive disorders of pregnancy are the third leading cause of maternal death in the United States. Hypertensive disorders of pregnancy, including preeclampsia, lead to preterm delivery, morbidity and mortality of mother, fetus, and neonate, and are a predictor of development of chronic maternal hypertension, cardiovascular disease, and renal disease. Maternal obesity is increasing dramatically in the patient population, and is an independent risk factor for hypertension and preeclampsia, increasing the risk by two- to four-fold. To date, no effective preventative measure has been found to reduce the risk of preeclampsia or hypertension in high risk pregnant patients. However, observational studies have shown that patients who exercise or who have increased physical activity before and during pregnancy have lower rates of preeclampsia, hypertension, and gestational diabetes. Exercise has been shown in numerous studies to be safe in pregnancy, and is recommended by the American College of Obstetrics and Gynecology as part of routine prenatal care. However, aerobic exercise can be viewed by patients to be difficult to perform during pregnancy, particularly when the patient is obese and at later gestations. Adherence to exercise regimens is therefore low in this patient group. Dynamic resistance training has been shown to lower mean blood pressure both acutely and long term in non-pregnant hypertensive patients, and can be performed more easily by patients with mobility issues. This intervention has not been studied in an obese pregnant population for its effects on blood pressure throughout pregnancy.

The long term goal is to develop an intervention that will reduce the barriers to exercise of obese pregnant women that will, in turn, reduce their risk of developing preeclampsia and other hypertensive disorders of pregnancy. The specific objective of this proposal is to study the effect of a structured resistance training exercise intervention on blood pressure in obese pregnant woman, who would be considered high risk for development of hypertensive disorders based on pre-pregnancy BMI. The central hypothesis is that obese pregnant patients who participate in a regular, structured resistance training exercise regimen will have a decrease in mean arterial blood pressure compared to obese pregnant patients who are strongly encouraged to do aerobic exercise (lifestyle intervention) or who participate in routine prenatal care. The investigators formulated this hypothesis, in part, based upon previous studies found in the literature performed in non-pregnant hypertensive patients. The investigators will extrapolate from the experience and methods of the collaborators, who have studied the effects of exercise on gestational diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patient's BMI must be ≥ 30 and ≤ 40.
* Established viable singleton pregnancy <13 weeks

Exclusion Criteria:

* Multiple gestations.
* Maternal diabetes established pre-pregnancy by standard guidelines
* Congenital or acquired heart disease
* Use of antihypertensive medication
* Inability to exercise
* Restrictive lung disease
* History of shortened/incompetent cervix
* History of preterm labor

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2010-11; Primary Completion 2014-07 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in mean arterial blood pressure | <13 weeks gestation-postpartum visit

SECONDARY OUTCOMES:
Hypertension of pregnancy or preeclampsia
Gestational weight gain
Neonatal weight
Proteinuria
Serum markers for hypertension risk
Activity level
  Measured with activity logos
Number of steps per week
  Pedometer measurement
Weight retention at postpartum visit
Mode of delivery
  Vaginal versus cesarean

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States